CLINICAL TRIAL: NCT01799187
Title: Randomized Controlled Research of Revascularization in Immature Permanent Teeth With Periapical Periodontitis
Brief Title: Research of Revascularization in Immature Teeth With Periapical Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Junqi Ling (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor-Investigator, Junqi Ling, Dean, professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5010YT; jqling (Registry Identifier: Junqi Ling)
Record Dates: First submitted 2013-02-24; First posted 2013-02-26 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Periapical Periodontitis
Keywords: Immature Permanent Teeth
MeSH Terms: conditions — Periapical Periodontitis | interventions — Apexification

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- revascularization (Experimental): revascularization is is an alternative new treatment of immature permanent teeth with necrotic pulp. The use of triple antibiotic paste is followed by Induction of bleeding from the apical root during this intervention.
  Interventions: Procedure: revascularization
- apexification (Active Comparator): apexification is a traditional therapy of immature permanent teeth with necrotic pulp.calcium hydroxide is served as medication to induce the developing of root .
  Interventions: Procedure: apexification

INTERVENTIONS:
Procedure: revascularization — revascularization include 3 steps: root disinfected,induction of bleeding and revascularization include 3 steps: root disinfected,induction of bleeding and sealing
  Arms: revascularization
Procedure: apexification — apexification uses calcium hydroxide as root medication
  Arms: apexification

SUMMARY:
Revascularization is an alternative new treatment of immature permanent teeth with necrotic pulp nowadays while apexification is the traditional therapy. The investigators suppose that revascularization is superior to apexification at developing the root of immature permanent teeth and reducing the risk of root fracture,and the research is designed.

DETAILED DESCRIPTION:
The investigators design to collect a group of patients presenting immature permanent teeth with periapical periodontitis in certain criterion. The investigators will divide the patients into two groups randomly. One group will get treated with revascularization while the other with apexification. The investigators want to evaluate the short-term and long-term effects of the two groups to get a conclusion of the clinical value of revascularization.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of periapical periodontitis
* must be immature permanent teeth
* must be local Guangzhou

Exclusion Criteria:

* blood disease
* residual root that is advised to extract
* serious periodontitis
* women in pregnancy

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 190 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Evidence of lesion healing confirmed by cone beam computed tomography | one year

CONTACTS AND LOCATIONS:
Overall Officials: ling j qi, PhD, Study Chair — Guanghua hospital of stomotology,Sun Yat-sen University
Locations (1):
- Guanghua hospital of stomotology,Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Jung IY, Lee SJ, Hargreaves KM. Biologically based treatment of immature permanent teeth with pulpal necrosis: a case series. J Endod. 2008 Jul;34(7):876-87. doi: 10.1016/j.joen.2008.03.023. Epub 2008 May 16. PMID 18571000